CLINICAL TRIAL: NCT03598465
Title: Evaluating the Association Between Sphingolipid Metabolites and Post-hepatectomy Liver Failure
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2018-033
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Post-hepatectomy Liver Failure
Keywords: Post-hepatectomy liver failure; Sphingolipids metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHLF Group: The investigators will define PHLF as a postoperatively acquired deterioration in synthetic, excretory, and detoxifying functions of liver. According to the PHLF definition and grading criteria established by International Liver Group of Liver Surgery (ISGLS) in 2011 (Surgery,2011,149(5):713-724), PHLF will be diagnosed by an increased PT-INR and concomitant hyperbilirubinemia on or after postoperative day 5.
- Non-PHLF Group: Non-PHLF will be defined as normal liver function in terms of normal PT-INR and bilirubin levels after hepatectomy on or after postoperative day 5.

SUMMARY:
Hepatectomy is an essential treatment for various benign and malignant diseases of the liver. However, post-hepatectomy liver failure (PHLF) is still a life-threatening complication after hepatectomy. The pathophysiological mechanism of PHLF has not yet been fully elucidated, and there is still a lack of effective strategies for either prevention or therapy of PHLF.

Sphingolipids include ceramides (CER), sphingomyelins (SM), glycosphingolipids (GSL), sphingosine (SPH), and sphingosine-1-phosphate (S1P) are multi-functional lipids that regulates cell proliferation, cell survival, cell death, inflammation, tissue fibrosis, cancer cell metastasis, and invasion. Liver is a main organ for metabolizing sphingolipids, dysregulation of specific sphingolipids is associated with several liver diseases, therefore sphingolipids have been proposed to be biomarkers of liver diseases, including hepatitis, liver cancer, fatty liver diseases, and liver fibrosis. Moreover, several studies have shown CER, SPH and S1P are critical in regulating pathophysiology of liver diseases, including liver regeneration, necrosis, and inflammation. Given that PHLF causes dramatic dysregulation in biochemical metabolism in liver, the investigators hypothesize that dysregulation of sphingolipid metabolism may also occur in PHLF, and the dysregulation of specific sphingolipids may serve as a biomarker or regulator during progression and recovery of PHLF.

This project will examine the association between sphingolipid metabolism and PHLF. Levels of sphingolipid metabolites and their related enzymes in plasma and liver tissue of patients with hepatic resection will be measured by using liquid chromatograph/electrospray ionization/mass spectrometry (LC-ESI-MS/MS) and high-throughput real-time quantitative PCR. This project will facilitate us to identify specific sphingolipid metabolites as biomarker and regulator of PHLF.

DETAILED DESCRIPTION:
Liver resection is an effective treatment for both benign and malignant liver diseases. However, post-hepatectomy liver failure (PHLF) is still a life-threatening complication of liver resection. The pathophysiological mechanism of PHLF has not yet been fully studied, and there is still a lack of effective strategies for either prevention or therapy of PHLF. The investigation on PHLF has important clinical significance.

Sphingolipids are a group of bioactive lipids, including ceramides (CER), sphingomyelins (SM), glycosphingolipids (GSL), etc. CER are the basic structure that constitute sphingolipids. CER are composed of long-chain bases of sphingosine and different fatty acid carbon chains. CER are of various species. According to the saturation of fatty acid carbon chains, CER can be divided into saturated CER and unsaturated CER. CER can be divided into four species, including short chain (less than 6 carbon atoms), medium chain (6-12 carbon atoms), long chain (14-20 carbon atoms), and super long chain (more than 22 carbon atoms) . Pathways of CER generation include de novo synthesis, complex sphingolipid lipid degradation pathways, and salvage synthesis pathways. CER are degraded to produce sphingosine (SPH), which can be phosphorylated to produce S1P. CER and its metabolites SPH and S1P are enigmatic lipids that regulates cell survival, death, inflammation, tissue fibrosis, cancer metastasis, and cancer invasion. Hepatocytes express activities of various sphingolipid enzymes, which makes liver an important organ for sphingolipid metabolism. Emerging evidences have shown that dysregulation of sphingolipid metabolite are associated with development and progression of certain liver diseases. In animal studies, dysregulation of ceramides has been indicated in hepatocyte survival, liver injury, and liver failure. In clinical studies, dysregulation of specific ceramide species has been identified to be associated with decompensation of cirrhosis, liver fibrosis, hepatitis, hepatocellular carcinoma. In the light of these evidences, the investigators hypothesize that dysregulation of sphingolipid metabolism may be associated with PHLF.

The investigators have established a quantitative method to measure different types of sphingolipids in human plasma, tissues, and cells using liquid chromatograph/electrospray ionization/mass spectrometry (LC-ESI-MS/MS), including C12-CER, C16-CER, C18-CER, C18:1-CER, C20-CER, C22-CER, C24-CER, C24:1-CER, SPH, S1P, C12-SM, C12-LacCER, C12-GluCER. In order to examine the correlation between sphingolipid metabolism and PHLF, the investigators will collect plasma of patients during peri-operation period of hepatectomy, after lipid extraction, the levels of sphingolipids will be measured by LC-ESI-MS/MS technology. Moreover, expression of sphingolipid-metabolizing enzymes in liver issues will be determined using high-throughput real-time quantitative PCR. The diagnostic criteria and grading of PHLF will be performed following criteria of International Liver Group of Liver Surgery. In the end, the investigators will analyze the correlation between sphingolipid metabolites and PHLF. This project will facilitate us to identify specific sphingolipid metabolites as biomarker and regulator of PHLF, and shed the light on the study of PHLF prevention and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepts hepatectomy
* In case of liver cancer, patient should received radical resection of R0 standards.

Exclusion criteria：

* Liver cancer invaded portal vein, common hepatic duct, hepatic vein trunk and/or inferior vena cava. Or the presence of extrahepatic metastases.
* Biliary obstruction, or surgery with exploration and reconstruction of bile duct.
* Surgery with splenectomy or splenic artery ligation.
* Patients with significant heart, lung, kidney and other organs of major diseases before surgery.
* The patients died in 90 days after surgery except for PHLF.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients who receive hepatectomy for benign or malignant disease in the department of Hepatobiliary Surgery of Nanfang Hospital Southern Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Post-hepatectomy liver failure (PHLF) | On or after postoperative day 5 of hepatectomy.
  Liver failure caused by hepatectomy. (Surgery,2011,149(5):713-724).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhou, MD., Study Director — Nanfang Hospital, Southern Medical University; Kai Wang, MD.PhD., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (3):
- China (3):
  - The first people's hospital of Foshan, Foshan, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The second people's hospital of Shenzhen, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Derived] Liang H, Liu H, Li J, Wang B, Huang P, Guo W, Zhuang B, Liao L, Li Q, Wu X, Peng T, Lai Z, Tang S, Zhu B, Gao J, Lin S, Huang C, Liu C, Zeng M, Qian J, Zhang Q, Zhou J, Deng X, Li C, Wang K. Prospective multicenter validation of preoperative plasma ceramides as novel predictive biomarkers for clinically relevant post-hepatectomy liver failure. Int J Surg. 2025 Oct 1;111(10):6843-6856. doi: 10.1097/JS9.0000000000002791. Epub 2025 Jun 24. PMID 40557443
- See also: The definition and diagnostic criteria of post-hepatectomy liver failure were proposed by International Liver Group of Liver Surgery(ISGLS) in 2011. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Posthepatectomy+liver+failure%3A+A+definition+and+grading+by+the+International+Study+Group+of+Liver+Surgerywww.ncbi.nlm.nih.gov/pubmed/?term=Posthepatectomy+liver+failure%3A+A+definition+and+grading+by+the+International+Study+Group+of+Liver+Surgerywww.ncbi.nlm.nih.gov/pubmed/?term=Posthepatectomy+liver+failure%3A+A+definition+and+grading+by+the+International+Study+Group+of+Liver+Surgerywww.ncbi.nlm.nih.gov/pubmed/?term=Posthepatectomy+liver+failure%3A+A+definition+and+grading+by+the+International+Study+Group+of+Liver+Surgerywww.ncbi.nlm.nih.gov/pubmed/?term=Posthepatectomy+liver+failure%3A+A+definition+and+grading+by+the+International+Study+Group+of+Liver+Surgerywww.ncbi.nlm.nih.gov/pubmed/?term=Posthepatectomy+liver+failure%3A+A+definition+and+grading+by+the+International+Study+Group+of+Liver+Surgery

DOCUMENTS (1):
  • Informed Consent Form (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT03598465/ICF_000.pdf